CLINICAL TRIAL: NCT04191564
Title: Impact of Low Perfusion by High Intraabdominal Pressure and Low Blood Pressure on Stapling Quality Measured as Thickness Difference Between Staples and Stomach Wall and by Bursting Pressure of Excluded Stomach
Brief Title: Effect of Anesthetic Conditions on Stapling Thickness and Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Jan Mulier, Principal investigator, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020RCTStaplingcondition
Record Dates: First submitted 2019-12-01; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Gastrectomy

STUDY DESIGN:
Intervention Model Description: low perfusion
Masking Description: normal perfusion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low perfusion (Experimental): fluid restriction based on the goal directed fluid therapy is maintained during the whole case and a state of low perfusion is created by reducing the systolic blood pressure below 100 mmHg by vasoactive medications like cleviprex or nicardipine, by increasing positive end expiratory pressure (PEEP) and by a very short period of a high IAP of 20 mmHg only during firing.
  Interventions: Procedure: low perfusion state
- normal perfusion (Experimental): Perfusion pressure is maintained above 100 mmHg with free fluid loading iv and the lowest IAP possible during the whole procedure.
  Interventions: Procedure: normal perfusion state

INTERVENTIONS:
Procedure: low perfusion state — reduce SAP below 100 mmHg
  Arms: low perfusion
Procedure: normal perfusion state — maintain SAP above 100 mmHg
  Arms: normal perfusion

SUMMARY:
the excluded stomach during sleeve gastrectomy can be investigated post removal outside the patient. During stapling it is common to reduce systolic arterial blood pressure (SAP) below 100 mmHg to reduce peritoneal perfusion and have better compression. Higher intra abdominal pressures reduce also the peritoneal and mucosal perfusion and might help to improve stapling compression. Stapling compression can be evaluated by measuring stapling thickness and compare it with stomach wall thickness or by measuring leaks during leak test or better outside the patient on the excised stomach with a bursting pressure.

DETAILED DESCRIPTION:
Patients are randomized to two groups: group standard perfusion means that the SAP is kept between 100 and 140 mmHg by adapting depth of anesthesia, by level of post expiratory pressure or by giving vasoconstriction.

low perfusion group means that

1. systolic blood pressure is kept below 100 mmHg from the first linear staple till the last by using a Clevidipine infusion to regulate the blood pressure accurate just below 100 mmHg for a short time while needed.
2. goal directed fluid therapy using 100 ml/h fluid intravenous and extra load of fluid if pulse pressure variation > 20 %
3. increase intra abdominal pressure (IAP) up to 20 mmHg inly during stapling and return to minimum IAP needed to achieve 3 liter workspace.

The resected stomach is removed and analyzed outside the body before throwing away:

ELIGIBILITY:
Inclusion Criteria:

* primary sleeve gastrectomy

Exclusion Criteria:

* allergy to one of the drugs used intra operative
* liver, renal, cardiac or lung disease with limited function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
staple thickness in mm | on excised stomach before being discarded within 1 hour after surgery
  each staple is measured with thickness monitor
stomach thickness in mm close to staple measurement | on excised stomach before being discarded within 1 hour after surgery
  with a constant pressure thickness is measured every 10 seconds till 1 minute
bursting pressure in mmHg | on excised stomach before being discarded within 1 hour after surgery
  excised stomach is inflated with air under water with increasing pressure that is recorded. At moment of first bubbles intra gastric pressure is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jan Paul Mulier, Principal Investigator — AZSint Jan AV
Locations (1):
- Azsintjan, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No